CLINICAL TRIAL: NCT01283542
Title: An Open-Label, Single Arm, Phase II Study to Evaluate the Efficacy and Safety of Pasireotide LAR on the Treatment of Patients With Clinically Non-Functioning Pituitary Adenoma
Brief Title: Evaluate the Efficacy and Safety of Pasireotide LAR (Long Acting Release) on the Treatment of Patients With Clinically Non-Functioning Pituitary Adenoma.
Acronym: Passion I
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSOM230D2401
Record Dates: First submitted 2010-12-17; First posted 2011-01-26 (Estimated); Results first posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Non-functioning Pituitary Adenoma
Keywords: Non-functioning pituitary adenoma,; pasireotide LAR,; tumor volume

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pasireotide LAR (Experimental): All patients will receive pasireotide LAR (long acting release) 60 mg every 28 ± 3 days for 24 weeks
  Interventions: Drug: Pasireotide LAR

INTERVENTIONS:
Drug: Pasireotide LAR — 20 and 40 mg of powder in vials and 2 mL of vehicle in ampoules (for reconstitution) administered as a depot intragluteal IM (intramuscular) injection

SUMMARY:
This study assessed pasireotide LAR efficacy on patients with non-functioning pituitary adenomas concerning tumor growth.

ELIGIBILITY:
Inclusion Criteria:

* Non-functioning pituitary adenoma ≥ 1cm, patients without any previous treatment for the tumor
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1

Exclusion Criteria:

* Patients who required a surgical intervention for relief of any sign or symptom associated with tumor compression
* Previous pituitary surgery
* Previous medical treatment for pituitary tumor
* Patients who had received pituitary irradiation within 10 years prior to randomization
* Prolactin (PRL) levels > 100 ng/mL. PRL evaluation should have been performed with diluted samples to ensure "hook effect." was avoided
* Patients who presented prolactinomas, acromegaly or Cushing's disease
* Patients with compression of the optic chiasm causing acute clinically significant visual field defects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-11-26 (Actual); Primary Completion 2017-09-12 (Actual); Study Completion 2017-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- Brazil (6):
  - Novartis Investigative Site, Fortaleza, Ceará
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Joinville, Santa Catarina
  - Novartis Investigative Site, Botucatu, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty seven patients were screened and 21 met eligibility requirements.
Period: Main Phase
Arm/Group | Pasireotide LAR
Started | 20
Full Analysis Set (FAS) (received at least 1 dose of study medication) | 20
Safety Analysis Set (rec'd at least 1 dose of drug + 1 at least one post-BL safety assessment) | 20
Completed | 13
Not Completed | 7
Not completed — Acute or progressive vision loss | 1
Not completed — Uncontrolled diabetes mellitus | 1
Not completed — abnormal laboratory values | 5
Period: Extension Phase
Arm/Group | Pasireotide LAR
Started | 13
Full Analysis Set (FAS) (received at least 1 dose of study drug) | 13
Safety Analysis Set (rec'd at least 1 dose of drug + 1 at least one post-BL safety assessment) | 13
Completed | 10
Not Completed | 3
Not completed — Physician Decision | 1
Not completed — Adverse Event | 1
Not completed — Administrative problems | 1

BASELINE CHARACTERISTICS:
Population: Baseline participants met eligibility requirements and received at least 1 dose of study medication
Arm/Group | Pasireotide LAR
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.65 (11.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian ancestry | 13
  Black/African ancestry | 5
  Asian ancestry | 1
  Other | 1
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 26.95 (4.53)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Non-functioning Pituitary Adenomas (NFPA) Who Achieve Tumor Volume Reduction of at Least 20% After 24 Weeks (FAS)
Description: Tumor volume was evaluated by MRI. MRIs were performed and processed according to the guidelines of the central evaluator's facility.The pituitary adenomas were measured by a neuro-radiologist, using manual tracing together with the imaging analysis software. The largest diameter at any plan determined the maximum diameter of the tumor. A change ≥ 20% in the original volume of the tumor was considered to be clinically significant. Evaluable participants required tumor volume assessment at baseline and at week 24.
Time Frame: Baseline up to 24 weeks
Population: Evaluable participants required tumor volume assessment at baseline and at week 24
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pasireotide LAR
Number analyzed (Participants) | 12
percentage of participants | 16.7 [2.1 to 48.4]

2. Secondary Outcome: Tumor Volume Main Phase (FAS)
Description: Tumor volume was evaluated by MRI. MRIs were performed and processed according to the guidelines of the central evaluator's facility. The pituitary adenomas were measured by a neuro-radiologist, using manual tracing together with the imaging analysis software. The largest diameter at any plan determined the maximum diameter of the tumor.
Time Frame: baseline to week 4, 12, 24
Population: number of participants with evaluable data varied across visits
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Pasireotide LAR
Number analyzed (Participants) | 20
cm^3
  Main Baseline | 2.97 (2.53)
  Main Week 4 | 4.31 (6.66)
  Main Week 12: number analyzed (Participants) | 19
  Main Week 12 | 4.31 (6.66)
  Main Week 24 | 3.39 (3.15)

3. Secondary Outcome: Tumor Volume in Extension Phase (FAS)
Description: as for outcome 2
Time Frame: baseline to week 48, 72, 96
Population: number of participants with evaluable data varied across visits
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Pasireotide LAR
Number analyzed (Participants) | 13
cm^3
  Extension Week 48 | 3.57 (3.25)
  Extension Week 72 | 3.12 (2.48)
  Extension Week 96 | 1.70 (1.02)

4. Secondary Outcome: Tumor Volume Change From Baseline in Main Phase (FAS)
Description: as for outcome 2
Time Frame: baseline to week 4, 12, 24
Population: number of participants with evaluable data varied across visits
Measure: Mean (95% Confidence Interval); unit: cm^3
Arm/Group | Pasireotide LAR
Number analyzed (Participants) | 20
cm^3
  Main Week 4 | 1.25 [-1.70 to 4.20]
  Main Week 12: number analyzed (Participants) | 19
  Main Week 12 | 0.66 [-0.45 to 1.76]
  Main Week 24 | 0.23 [-1.24 to 1.71]

5. Secondary Outcome: Tumor Volume Change From Baseline in Extension Phase (FAS)
Description: as for outcome 2
Time Frame: baseline to week 48, 72, 96
Population: number of participants with evaluable data varied across visits
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Pasireotide LAR
Number analyzed (Participants) | 13
cm^3
  Extension Week 48 | 0.53 (2.19)
  Extension Week 72: number analyzed (Participants) | 12
  Extension Week 72 | -0.14 (0.63)
  Extension Week 96: number analyzed (Participants) | 11
  Extension Week 96 | 0.0 (0.90)

6. Secondary Outcome: Tumor Volume Percent Change From Baseline in Main Phase (FAS)
Description: as for outcome 2
Time Frame: baseline to week 4, 12, 24
Population: number of participants with evaluable data varied across visits
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Pasireotide LAR
Number analyzed (Participants) | 20
percent change
  Main Week 4 | 36.92 [-52.11 to 125.94]
  Main Week 12: number analyzed (Participants) | 19
  Main Week 12 | 39.36 [-42.19 to 120.91]
  Main Week 24 | 7.98 [-32.79 to 48.74]

7. Secondary Outcome: Tumor Volume Percent Change From Baseline in Extension Phase (FAS)
Description: as for outcome 2
Time Frame: baseline to week 48, 72, 96
Population: number of participants with evaluable data varied across visits
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Pasireotide LAR
Number analyzed (Participants) | 13
percent change
  Extension Week 48 | 14.83 (67.28)
  Extension Week 72: number analyzed (Participants) | 12
  Extension Week 72 | -2.57 (14.33)
  Extension Week 96: number analyzed (Participants) | 11
  Extension Week 96 | -1.59 (53.09)

8. Secondary Outcome: Percentage of Patients Achieving Tumour Volume Reduction in Main Phase (FAS)
Description: as for outcome 2
Time Frame: baseline to week 4, 12, 24
Population: number of participants with evaluable data varied across visits
Measure: Number; unit: percentage of patients
Arm/Group | Pasireotide LAR
Number analyzed (Participants) | 20
percentage of patients
  Week 4: number analyzed (Participants) | 19
  Week 4 | 47.4
  Week 12: number analyzed (Participants) | 17
  Week 12 | 41.2
  Week 24: number analyzed (Participants) | 12
  Week 24 | 75.0

9. Secondary Outcome: Percentage of Patients Achieving Tumour Volume Reduction of at Least ≥ 20% in Main Phase (FAS)
Description: as for outcome 2
Time Frame: baseline to week 4, 12, 24
Population: number of participants with evaluable data varied across visits
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Pasireotide LAR
Number analyzed (Participants) | 20
percentage of patients
  Main Week 4: number analyzed (Participants) | 19
  Main Week 4 | 10.5 [1.3 to 33.1]
  Main Week 12: number analyzed (Participants) | 17
  Main Week 12 | 5.9 [0.1 to 28.7]
  Main Week 24: number analyzed (Participants) | 12
  Main Week 24 | 16.7 [2.1 to 48.4]

10. Secondary Outcome: Percentage of Patients Achieving Tumour Volume Reduction in Extension Phase (FAS)
Description: as for outcome 2
Time Frame: baseline to week 48, 72, 96
Population: number of participants with evaluable data varied across visits
Measure: Number; unit: percentage of patients
Arm/Group | Pasireotide LAR
Number analyzed (Participants) | 13
percentage of patients
  Extension Week 48: number analyzed (Participants) | 10
  Extension Week 48 | 10.0
  Extension Week 72: number analyzed (Participants) | 8
  Extension Week 72 | 12.5
  Extension Week 96: number analyzed (Participants) | 2
  Extension Week 96 | 50.0

11. Secondary Outcome: Percentage of Patients Achieving Tumour Volume Reduction of at Least ≥ 20% in Extension Phase (FAS)
Description: as for outcome 2
Time Frame: baseline to week 48, 72, 96
Population: number of participants with evaluable data varied across visits
Measure: Number; unit: percentage of patients
Arm/Group | Pasireotide LAR
Number analyzed (Participants) | 13
percentage of patients
  Extension Week 48: number analyzed (Participants) | 10
  Extension Week 48 | 10.0
  Extension Week 72: number analyzed (Participants) | 8
  Extension Week 72 | 12.5
  Extension Week 96: number analyzed (Participants) | 2
  Extension Week 96 | 50.0

12. Secondary Outcome: Percentage of Participants Reporting Absence and Presence of Relevant Disease-related Symptoms (FAS)
Description: The absence and presence of disease-related symptoms were reported by patients and recorded by the medical staff. Patients classified the symptoms according to a 5-point scale (0 = absent, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe
Time Frame: Baseline and at weeks 4, 12,24,48,72, 96
Population: number of participants varied across visits
Measure: Number; unit: percentage of participants
Groups:
- Baseline: Baseline of Main Phase
- Week 4: Week 4 of Main Phase
- Week 12: Week 12 of Main Phase
- Week 24: Week 24 of Main Phase
- Week 48: Week 48 of Extension Phase
- Week 72: Week 72 of Extension Phase
- Week 96: Week 96 of Extension Phase
Arm/Group | Baseline | Week 4 | Week 12 | Week 24 | Week 48 | Week 72 | Week 96
Number analyzed (Participants) | 20 | 20 | 19 | 20 | 13 | 12 | 11
percentage of participants
  Headache Absent | 45.0 | 75.0 | 52.6 | 45.0 | 61.5 | 58.3 | 70.0
  Headache Mild | 30.0 | 10.0 | 36.8 | 45.0 | 7.7 | 8.3 | 0.0
  Headache Moderate | 25.0 | 15.0 | 10.5 | 10.0 | 30.8 | 33.3 | 20.0
  Headache Severe | 0 | 0 | 0 | 0 | 0 | 0 | 10.0
  Visual Disturbances Absent | 80.0 | 80.0 | 84.2 | 85.0 | 76.9 | 83.3 | 80.0
  Visual Disturbances Mild | 10.0 | 10.0 | 10.5 | 10.0 | 7.7 | 0 | 0
  Visual Disturbances Moderate | 5.0 | 5.0 | 5.3 | 5.0 | 15.4 | 16.7 | 20.0
  Visual Disturbances Severe | 5.0 | 5.0 | 0 | 0 | 0 | 0 | 0
  Fatigue Absent | 80.0 | 80.0 | 73.7 | 75.0 | 69.2 | 58.3 | 70.0
  Fatigue Mild | 15.0 | 15.0 | 21.1 | 20.0 | 30.8 | 33.3 | 30.0
  Fatigue Moderate | 5.0 | 0 | 5.3 | 5.0 | 0 | 8.3 | 0
  Fatigue Severe | 0 | 5.0 | 0 | 0 | 0 | 0 | 0
  Decreased libido Absent | 55.0 | 65.0 | 68.4 | 65.0 | 61.5 | 66.7 | 70.0
  Decreased libido Mild | 10.0 | 10.0 | 10.5 | 10.0 | 23.1 | 25.0 | 0
  Decreased libido Moderate | 20.0 | 10.0 | 5.3 | 10.0 | 0 | 0 | 20.0
  Decreased libido Severe | 5.0 | 15.0 | 15.8 | 15.0 | 15.4 | 8.3 | 10.0
  Decreased libido Very severe | 10.0 | 0 | 0 | 0 | 0 | 0 | 0
  Erectile dysfunction Yes | 22.2 | 11.1 | 11.1 | 11.1 | 0 | 0 | 0
  Erectile dysfunction No | 77.8 | 88.9 | 88.9 | 88.9 | 100.0 | 100.0 | 100.0
  Regular Menses Yes | 45.5 | 55.6 | 62.5 | 55.6 | 60.0 | 50.0 | 50.0
  Regular Menses No | 54.5 | 44.4 | 37.5 | 44.4 | 40.0 | 50.0 | 50.0

13. Secondary Outcome: Mean GH and IGF-1 Hormone Levels During Main and Extension Phases (FAS)
Description: Hormone levels, including those of GH, IGF-1, and prolactin were evaluated by a central lab
Time Frame: Baseline and at weeks 24, 48, 96
Population: number of participants with evaluable data varied across visits
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Baseline | Week 24 | Week 48 | Week 96
Number analyzed (Participants) | 20 | 20 | 13 | 11
ng/mL
  GH: number analyzed (Participants) | 19 | 17 | 12 | 9
  GH | 0.31 (0.63) | 1.11 (4.10) | 0.15 (0.15) | 0.12 (0.07)
  IGF-1: number analyzed (Participants) | 17 | 15 | 12 | 9
  IGF-1 | 130.73 (44.4) | 72.59 (35.55) | 66.23 (31.46) | 70.82 (32.67)
  Prolactin: number analyzed (Participants) | 20 | 16 | 12 | 10
  Prolactin | 16.90 (12.91) | 13.89 (17.32) | 9.03 (6.27) | 7.62 (8.33)

14. Secondary Outcome: Mean ACTH and Estradiol Hormone Levels During Main and Extension Phases (FAS)
Description: Hormone levels, including those of growth hormone (GH),insulin-like growth factor 1 (IGF-1), follicle-stimulating hormone (FSH), luteinizing hormone (LH), adrenocorticotropic hormone (ACTH), thyroid-stimulating hormone (TSH), prolactin, cortisol, free thyroxine (free T4), and estradiol (for women) or testosterone (for men), were evaluated by a central lab
Time Frame: Baseline and at weeks 24, 48, 96
Population: participants with evaluable data varied across visits
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Baseline | Week 24 | Week 48 | Week 96
Number analyzed (Participants) | 20 | 20 | 13 | 11
pg/mL
  ACTH: number analyzed (Participants) | 14 | 16 | 9 | 10
  ACTH | 28.91 (37.07) | 23.18 (31.67) | 36.06 (33.09) | 29.90 (26.83)
  Estradiol: number analyzed (Participants) | 11 | 10 | 7 | 7
  Estradiol | 35.72 (21.03) | 32.12 (17.71) | 34.69 (14.74) | 19.98 (15.78)

15. Secondary Outcome: Mean Cortisol Hormone Levels During Main and Extension Phases (FAS)
Description: Hormone levels, including those of GH, IGF-1, follicle-stimulating hormone (FSH), luteinizing hormone (LH), adrenocorticotropic hormone (ACTH), thyroid-stimulating hormone (TSH), prolactin, cortisol, free T4, and estradiol (for women) or testosterone (for men), were evaluated by a central lab
Time Frame: Baseline and at weeks 24, 48, 96
Population: number participants with evaluable data varied across visits
Measure: Mean (Standard Deviation); unit: µg/dL
Arm/Group | Baseline | Week 24 | Week 48 | Week 96
Number analyzed (Participants) | 20 | 20 | 13 | 11
µg/dL | 12.60 (4.37) | 16.41 (8.28) | 12.12 (4.43) | 10.09 (3.12)

16. Secondary Outcome: Mean LH and FSH Hormone Levels During Main and Extension Phases (FAS)
Description: as for outcome 15
Time Frame: Baseline and at weeks 24, 48, 96
Population: participants with evaluable data varied across visits
Measure: Mean (Standard Deviation); unit: mUI/mL
Arm/Group | Baseline | Week 24 | Week 48 | Week 96
Number analyzed (Participants) | 20 | 20 | 13 | 11
mUI/mL
  LH: number analyzed (Participants) | 19 | 18 | 11 | 10
  LH | 5.57 (6.91) | 5.32 (7.25) | 7.44 (7.07) | 9.95 (9.56)
  FSH: number analyzed (Participants) | 19 | 17 | 12 | 10
  FSH | 11.83 (18.89) | 12.90 (20.00) | 16.23 (20.97) | 21.45 (24.56)

17. Secondary Outcome: Mean Testosterone and Free T4 Hormone Levels During Main and Extension Phases (FAS)
Description: as for outcome 15
Time Frame: Baseline and at weeks 24, 48, 96
Population: participants with evaluable data varied across visits
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Baseline | Week 24 | Week 48 | Week 96
Number analyzed (Participants) | 20 | 20 | 13 | 11
ng/dL
  Testosterone: number analyzed (Participants) | 8 | 5 | 5 | 7
  Testosterone | 452.21 (214.52) | 372.72 (205.25) | 517.52 (200.64) | 382.10 (179.79)
  Free T4: number analyzed (Participants) | 18 | 17 | 12 | 10
  Free T4 | 1.07 (0.12) | 1.13 (0.18) | 1.17 (0.17) | 1.04 (0.25)

18. Secondary Outcome: Mean TSH Hormone Levels During Main and Extension Phases (FAS)
Description: as for outcome 15
Time Frame: Baseline and at weeks 24, 48, 96
Population: participants with evaluable data varied across visits
Measure: Mean (Standard Deviation); unit: µUI/mL
Arm/Group | Baseline | Week 24 | Week 48 | Week 96
Number analyzed (Participants) | 20 | 20 | 13 | 11
µUI/mL | 151.81 (655.82) | 149.92 (628.93) | 1.67 (1.27) | 1.70 (1.33)

19. Secondary Outcome: Mean Alpha Subunit Levels in Main and Extension Phases (FAS)
Time Frame: Baseline and at weeks 12,24,48,72, 96
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Baseline | Week 12 | Week 24 | Week 48 | Week 72 | Week 96
Number analyzed (Participants) | 16 | 14 | 15 | 13 | 12 | 11
ng/mL | 242.27 (286.90) | 309.04 (270.52) | 192.11 (201.25) | 234.21 (182.59) | 286.78 (288.62) | 435.00 (310.87)

20. Secondary Outcome: Percentage of Participants With Reduction From Baseline of Alpha Subunit ≥50% in Main and Extension Phases (FAS)
Description: Alpha subunit levels were determined at a central laboratory.
Time Frame: Baseline up to approximately Week 96
Population: Evaluable participants had to have 50% reduction
Measure: Number; unit: percentage of participants
Arm/Group | Week 12 | Week 24 | Week 48 | Week 72 | Week 96
Number analyzed (Participants) | 14 | 15 | 10 | 10 | 6
percentage of participants | 8.3 | 28.6 | 12.5 | 22.2 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to approximately 104 weeks
Arm/Group | Pasireotide LAR
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 2/20
Other Adverse Events (participants affected / at risk) | 17/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pasireotide LAR (N=20)
Cholelithiasis (Hepatobiliary disorders) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pasireotide LAR (N=20)
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 5
Blood glucose increased (Investigations) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 5
Dyslipidaemia (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 9
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2012-03-26): https://cdn.clinicaltrials.gov/large-docs/42/NCT01283542/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-14): https://cdn.clinicaltrials.gov/large-docs/42/NCT01283542/SAP_001.pdf